CLINICAL TRIAL: NCT06602323
Title: Phase II Study of Total Marrow and Lymphoid Irradiation (TMLI) Administered in Combination With a Reduced-intensity Regimen Based on Fludarabine and Melphalan as Conditioning for Allogeneic Hematopoietic Stem Cell Transplantation (AHSCT) in Patients With High Risk Myelodysplastic Syndrome or Acute Myeloid Leukemia.
Brief Title: TMLI/Fludarabine/Melphalan Conditioning for Allogeneic Transplantation in High-risk Myelodysplastic Syndrome or Acute Myeloid Leukemia.
Acronym: TMLI-RI
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TMLI-RI; 2024-514483-11-00 (EU CTIS Number)
Record Dates: First submitted 2024-09-16; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Myelodysplastic Syndromes; Acute Myeloid Leukemia
Keywords: Myelodysplastic Syndromes; Acute Myeloid Leukemia
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute

STUDY DESIGN:
Intervention Model Description: A 3+3 de-escalation design comprising a patient safety-lead phase will be applied in successive patient cohorts:
  Initially, 3 patients will be treated at the starting TMLI dose (Dose Level 1, 1200 cGy). If 0 or 1 dose-limiting toxicity is observed among the first 6 patients at Dose Level 1, then 28 additional patients will be treated at this dose level (allowing for the evaluation of 34 patients treated at the target dose level). If ≥2/6 patients experience a dose-limiting toxicity at Dose Level 1, then the maximum tolerated dose has been exceeded and the next lower TMLI dose (Dose Level -1, 1100 cGy) will be expanded to up to 6 patients. If 0 or 1 patient out of 6 experiences a dose-limiting toxicity, this dose level will be further evaluated (n=28 additional patients). If ≥2/6 patients experience a dose-limiting toxicity, the next lower dose (Dose Level -2, 1000 cGy) level will be expanded applying the same criteria.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TMLI/Flu/Mel conditioning regimen (Single-arm) (Other): Single-arm.
  TMLI:
  Dose level 1: 1200 cGy = 150 cGy x 8 doses (liver, brain, and hepatic portal limited to 720 cGy) Dose level -1: 1100 cGy = 137.5 cGy x 8 doses (liver, brain, and hepatic portal limited to 720 cGy) Dose level -2: 1000 cGy = 125 cGy x 8 doses (liver, brain, and hepatic portal limited to 720 cGy) Dose levels above 1,200 cGy will not be considered in this protocol, as the dose to off-target avoidance organs would exceed the recommended levels in reduced-intensity transplants.
  TMLI will be administered by helical tomotherapy for 4 consecutive days (day -7 to day -4), delivering 2 fractions per day (a total of 8 doses) with a minimum of 6 hours between fractions.
  FLURADABINE:
  Dose: 25 mg/m2 Route of administration: intravenous. Treatment duration: for 4 consecutive days (day -7 to day -4 pre-transplant).
  MELPHALAN:
  Dose: 140 mg/m2 Route of administration: intravenous Treatment duration: for 1 day (day -2 pre-transplant).
  Interventions: Combination Product: TMLI/Flu/Mel

INTERVENTIONS:
Combination Product: TMLI/Flu/Mel — Targeted total bone marrow and lymphoid irradiation (TMLI) conformal therapy administered in combination with a reduced-intensity regimen based on Fludarabine and Melphalan.

SUMMARY:
The goal of this clinical trial is to learn if drugs (fludarabine and melphalan) combinated with a targeted irradiation (in bone marrow and in lymphoid tissue) works to treat blood cancers (high risk myelodysplastic syndrome or acute myeloid leukemia) in adults. It will also learn about the safety of this combination of drugs and irradiation. The main questions it aims to answer are:

* Does this combined therapy result in an improved survival and decreased relapse/progression rate after a bone marrow transplant?
* What toxicities or complications do participants have when taking this combined therapy?

Researchers will use this combined therapy to see if it works to treat high risk myelodysplastic syndrome or acute myeloid leukemia through the evaluation of the length of time (during the treatment and 2 years after the treatment) that a patient lives with the disease but it does not get worse (progression-free survival).

Participants will:

* Receive the combined therapy (study treatment) one week before the bone marrow transplant.
* Receive too post-transplant medication as per usual clinical practice.

Patients will have to attend medical visits (checkups and tests) for 2 years.

DETAILED DESCRIPTION:
This is a single-arm, single center phase II trial to evaluate the antileukemic activity and safety of the AHSCT TMLI/Flu/Mel conditioning regimen in patients with high-risk myelodysplastic syndrome or acute myeloid leukemia. A patient safety-lead phase will be carried out to ensure there are no unexpected toxicities. Ultimately, a total of 34 patients will be treated at the TMLI/Flu/Mel dose level deemed safe as determined during the introductory patient safety segment of this study.

Up to three dose levels can be studied. A 3+3 de-escalation design comprising a patient safety-lead phase will be applied in successive patient cohorts to evaluate the safety of the TMLI schedule and identify the optimal treatment dose:

Initially, 3 patients will be treated at the starting TMLI dose (Dose Level 1, 1200 cGy). If 0 or 1 DLT is observed among the first 6 patients at Dose Level 1, then 28 additional patients will be treated at this dose level (allowing for the evaluation of 34 patients treated at the target dose level). If ≥2/6 patients experience a DLT at Dose Level 1, then the MTD has been exceeded and the next lower TMLI dose (Dose Level -1, 1100 cGy) will be expanded to up to 6 patients. If 0 or 1 patient out of 6 experiences a DLT, this dose level will be further evaluated (n=28 additional patients). If ≥2/6 patients experience a DLT, the next lower dose (Dose Level -2, 1000 cGy) level will be expanded applying the same criteria. No further dose level reductions will be allowed beyond Dose Level -2.

No more than 3 patients may be <30 days after stem cell infusion at any time during patient safety introduction. The tacrolimus dose and MMF dose will remain fixed for all defined dose levels and will not be reduced at any time.

Considering this proposed design, the expected sample size of the study will be n=34 patients, with a potential minimum and maximum size of n=34 and n=46, respectively.

ELIGIBILITY:
Inclusion Criteria:

* The participant has the ability and willingness to sign the informed consent document. (For adults, only participants with mild cognitive abilities may use a legally authorized representative).
* Documented (signed) informed consent. The patient, family member, and doctor of the transplant staff (doctor, nurse, and social worker) meet at least once before the transplant procedure begins. During this meeting, all relevant information regarding the risks and benefits to the donor and recipient will be presented. Alternative treatment modalities will be discussed. The risks are explained in detail in the attached consent forms.
* Age: ≥ 50 years or Haematopoietic Cell Transplantation-Comorbidity Index pre-transplant score ≥ 3 or any other condition that precludes the use of a fully myeloablative conditioning regimen.
* Karnofsky's performance status ≥ 70%.
* Patients with myelodysplastic syndrome/acute myeloid leukemia or acute myeloid leukemia with relapsed/refractory active disease (i.e. ≥5% bone marrow blasts), or in complete remission or morphologic leukemia-free state with evidence of measurable residual disease as assessed by multiparameter flow cytometry (≥ 0,1%) or next-generation sequencing (in the case of fms-like tyrosine kinase-3 internal tandem duplication-mutated AML).
* All candidates for this study must have an 8/8 human leukocyte antigens-identical (A, B, C, DR) sibling donor or an unrelated donor with at least 8/8 human leukocyte antigens matching. A single allele mismatch in A, B, C, DR or dq and a kir mismatch in C shall be allowed. All combinations of donor/recipient "abo" blood types are acceptable; as even major "abo" compatibilities can be treated using a variety of techniques (red blood cell exchange or plasma exchange).
* The time elapsed since the end of the last induction or re-induction cycle must be greater than or equal to 14 days.
* Total bilirubin ≤ 1.5 mg/dL x Upper Limit of Normality OR 3 x upper limit of normal for Gilbert's disease.
* Serum glutamate oxaloacetate transaminase & serum glutamate pyruvate transaminase ≤ 5 x Upper Limit of Normality.
* Serum creatinine ≤ 1.3 mg/dL or creatinine clearance measured ≥ 80 mL/min for 24 hours of urine collection.
* Women of childbearing age only: Negative urine or serum pregnancy test.
* Men AND women of childbearing potential agree to use appropriate contraceptives (hormonal or barrier contraception or abstinence) prior to study entry and for six months following the duration of study participation. If a woman becomes pregnant or suspects she is pregnant while participating in the trial, she should inform her treating physician immediately.
* Pulmonary function tests: forced expiratory volume in one second (FEV1) and Carbon Monoxide Diffusion Capacity (DLCO) (adjusted for Hb) ≥ 50% from expected normal value.
* Patients should undergo cardiac evaluation with an electrocardiogram showing no ischemic changes or clinically relevant arrhythmia, and a ≥50% ejection fraction established by multigated acquisition scan or echocardiogram.
* ECG showing no ischemic changes or clinically significant arrhythmia.
* The time elapsed since the end of the last induction or reinduction cycle must be greater than or equal to 14 days.

Exclusion Criteria:

* Patients who have received a previous autologous (within the last year) or allogeneic transplant (at any time) are excluded.
* Previous radiation therapy which would preclude the use of TMLI.
* Plans during the trial to receive any other investigational (non-trial-related) agents.
* Uncontrolled disease, including ongoing or active infection.
* History of allergic reactions attributed to compounds of chemical or biological composition similar to cyclophosphamide or etoposide.
* Patients with other active malignancies are not eligible for this study, other than the malignancies discussed.
* Patients with a psychological or medical condition that the patient's physician deems unacceptable to proceed with allogeneic hematopoietic stem cell transplantation.
* Women who plan to become pregnant or breastfeed during the trial.
* Patients who do not agree to practice effective forms of contraception.
* Subjects who, in the opinion of the investigator, may not be able to meet the safety control requirements of the study.

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2028-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | From the start of therapy to 2 years after study treatment
  Time from the start of treatment to the date of death, disease relapse/progression, or date of last follow-up.

SECONDARY OUTCOMES:
Overall survival | From the start of therapy to 2 years after post-transplant.
  Quantification of time of patients who are still alive.
Cumulative incidence of recurrence/progression | From the start of therapy to 2 years after post-transplant.
  The event is relapse/progression either extramedullary or at bone marrow
Complete remission date | From the day of infusion to the day 30 post-transplant.
  The event is whether or not the patient has a documented complete remission.
Non-relapse mortality | From the start of therapy until 2 years after post-transplant.
  Number of deaths from causes other than relapse or progression.
Measurable residual disease | At 30, 90, 180 days and 1 year, 1.5 years and 2 years post-transplant.
  Measurable residual disease monitoring assessed by multiparameter flow cytometry.
Incidence of infection | 2 years after post-transplant.
  Microbiologically documented infections.
Adverse events | 2 years after post-transplant.
  Any untoward medical occurrence in a patient participating in clinical research that is associated in time with the use of a medicinal product, whether or not it is considered to be related to the investigational products.
Acute graft-versus-host disease grades 2-4 and 3-4 | 100 days post-transplant.
  This point is classified according to the NIH criteria.
Chronic graft-versus-host disease | 2 years after post-transplant.
  Chronic graft-versus-host disease is graded according to the NIH consensus staging.

CONTACTS AND LOCATIONS:
Overall Officials: José Antonio Pérez Simón, Hematologist, Principal Investigator — Hematology Department, Virgen del Rocío University Hospital, Seville)

IPD SHARING:
Plan to Share IPD: No